CLINICAL TRIAL: NCT02044042
Title: Mother-To-Child Transmission (MTCT) of Hepatitis C Virus and Spontaneous Viral Clearance in Infected Children: a Retrospective Study.
Brief Title: Vertical Transmission of Hepatitis C Virus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Stephane Mouly, MD PhD, Professor at University Paris VII Denis Diderot, physician, Hopital Lariboisière
Other Study IDs: Liver005
Record Dates: First submitted 2014-01-19; First posted 2014-01-23 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C; Transmission
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCV pregnant women: HCV chronically infected pregnant women, with a positive HCV RNA during pregnancy

SUMMARY:
Vertical HCV Transmission has been extensively studied, with a risk around 5% (range: 3 to 10%). Spontaneous viral clearance in infected children during childhood can occur, but data about this phenomenon are scarse, justifying the study.

DETAILED DESCRIPTION:
Hepatitis C Virus (HCV) Mother-To-Child Transmission (MTCT) has been extensively studied, with a risk around 5% (range: 3 to 10%) from chronically infected pregnant women with a positive HCV RNA during pregnancy. Risk factors include: HCV RNA load level, HIV-HCV co-infection, duration of labour, HCV genotype, child gender, and invasive procedures either during pregnancy or at birth. Hepatitis C Virus (HCV) Mother-To-Child Transmission (MTCT) mainly occurs during the last trimester of pregnancy or at birth or around the birth (El-Shabrawi et al., World Journal of Gastroenterology 2013). Currently, using caesarian section to reduce the risk of Hepatitis C Virus (HCV) Mother-To-Child Transmission (MTCT) is still debated and not recommended in International Guidelines (EASL 2012). Spontaneous viral clearance in infected children during childhood seems to occur in 20% of cases, with predisposing genetic factors (Ruiz-Extremera A et al. Hepatology 2011 ; 53 : 1830-1838) but data about this phenomenon are scarse (Rerksuppaphol S et al. J Gastroenterol Hepatol 2004), justifying the study.

ELIGIBILITY:
Inclusion Criteria:

* HCV chronically infected pregnant women
* with a positive HCV RNA
* who gave birth in the Maternity Department, Lariboisiere Hospital, Paris, France

Exclusion Criteria:

* negative HCV RNA during pregnancy
* acute HCV infection during pregnancy (previous negative HCV test during pregnancy)
* MTCT not to be tested (early child death for instance)

Ages: 9 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: HCV chronically infected pregnant women with a positive HCV RNA who gave birth in the Maternity Department, Lariboisiere Hospital, Paris, France
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
HCV status in children born from chronically HCV infected pregnant women | up to 10 years (expected average: 5 years)

SECONDARY OUTCOMES:
HCV RNA in children with positive HCV antibodies (Ab) | up to 10 years (expected average: 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre O SELLIER, M.D., Ph.D, Principal Investigator — Hopital Lariboisiere
Locations (1):
- Hopital Lariboisiere, Paris, France